CLINICAL TRIAL: NCT06951893
Title: Identification of Pre-surgical Phenotypic Indicators Predictive of Quality of Life Trajectories in Obese Patients Following Bariatric Surgery
Acronym: PHENOBEQOL73
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Metropole Savoie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHMS24006
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Obesity, Morbid; Obesity and Overweight; Bariatric Surgery; Bariatric Surgery Patients; Bariatric Surgery Patient; Bariatric Surgery (Sleeve Gastrectomy ); Bypass, Gastric
Keywords: GEROM73; PHENOBEQOL73
MeSH Terms: conditions — Obesity, Morbid; Obesity; Overweight | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone; Body Mass Index

STUDY DESIGN:
Intervention Model Description: each patient will complete questionary 6month before surgery, and then 12, 18 and 24 months after the surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- phenotype of patients during the GEROM73 program (Experimental): Anxiety, Depression, Eating disorders, Impact of Weight on Quality Of Life.Patients' weight, Body Mass index and Body schema
  Interventions: Other: Hospital Anxiety and Depression Scale; Other: Dutch Eating Behaviour Questionnary; Other: Impact of Weight on Quality Of Life; Other: body schema; Other: body mass index; Other: waist size

INTERVENTIONS:
Other: Hospital Anxiety and Depression Scale — It is a self-assessment questionnaire to identify the existence of anxious and depressive symptoms and to assess their severity.
Other: Dutch Eating Behaviour Questionnary — It allows the assessment of 3 distinct factors of eating behavior: cognitive restriction, emotional eating and externality. This tool was developed to better characterize the eating habits of obese subjects.
  10min
Other: Impact of Weight on Quality Of Life — The EQVOD is a validated French scale created from the Impact of Weight on Quality of Life (IWQOL) questionnaire. This self-administered questionnaire is specific to the sociocultural factors of obesity and its dietary treatment in France. The questionnaire is composed of five dimensions: physical impact (11 items), psychosocial impact (11 items), impact on sexual life (4 items), dietary well-being (5 items), and experience of diet/dietetics (5 items). The total number of items is 36.
Other: body schema — Tactile assessment of the body schema using a motorized caliper applied to different parts of the individual's body. The caliper is connected to a touch pad on which the person can report the difference felt between the two pressure points on their skin, using their thumb and index finger.
Other: body mass index — patient weighing at each visit
Other: waist size — waist size measure

SUMMARY:
This study aims to identify pre-operative phenotypic determinants predictive of quality of life trajectories in post-bariatric surgery patients. In addition, this study will have as a secondary objective the highlighting of a potential link between post-surgery quality of life trajectories and those of anxiety/depression scores, eating behaviors and body mass indices.

This study will be conducted during the usual care of patients undergoing the GEROM73 program, lasting a total of 30 months.

The GEROM73 program includes care for the six months preceding bariatric surgery and the 24 months following surgery. This program supports patients throughout their bariatric care..

Throughout the GEROM73 program, patients will complete questionnaires on anxiety, depression, eating disorders, Impact of Weight on Quality Of Life.

Patients' weight, body mass index and body schema will also be measured throughout the GEROM program.

ELIGIBILITY:
Inclusion Criteria:

* patient > 18years old
* Integrated into the GEROM73 surgical program and starting the intra-hospital program

Exclusion Criteria:

* Patients in a state of psychiatric decompensation
* Patients with cognitive disorders
* Patients with difficulties understanding the French language, spoken or written
* Pregnant, parturient, or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2030-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Time trajectories of EQVOD score during the 24 months post-surgery from measurements at M12, M18 and M24 according to phenotypic characteristics measured during the final pre-surgical assessment (M-1 of bariatric surgery) | one month befre surgery to 24 month post surgery
  Trajectory identification using latent class mixed models to classify patients into distinct EQVOD score trajectories over the 24 months post-surgery. The relationship between the 7 pre-surgery phenotypic characteristics and membership in the different trajectory classes will be tested in a multinomial logistic regression.

SECONDARY OUTCOMES:
quality of life trajectory groups defined by the analysis of the primary outcome measure, comparated to anxiety and depression measured at 12, 18 and 24 months. | 12, 18 and 24 month after surgery
  score of anxiety depression (HADS). The HAD (Hospital Anxiety and Depression Scale) assesses anxiety and depressive disorders (its use has been validated in French in the general population as well as in patients undergoing antidepressant treatment). This scale consists of 14 items rated from 0 to 3, of which 7 relate to anxiety and 7 to depression. Two scores are obtained and vary between 0 and 21.
  Interpretation takes into account two thresholds: the first, less than or equal to 7, corresponds to the absence of symptoms, and the second, greater than or equal to 11, indicates the presence of anxiety and/or depressive symptoms.
quality of life trajectory groups defined by the analysis of the primary outcome measure, comparated to Dutch Eating Behavior measured at 12, 18 and 24 months. | 12, 18 and 24 months after surgery
  Dutch Eating Behavior Questionnaire = DEBQ
  The Dutch Eating Behavior Questionnaire (DEBQ) is a 33-item self-report questionnaire developed by Van Strien et al. (1986), to assess three distinct eating behaviors in adults:
  1. emotional eating,
  2. external eating,
  3. restrained eating. Items on the DEBQ range from 1 (never) to 5 (very often), with higher scores indicating greater endorsement of the eating behavior.
quality of life trajectory groups defined by the analysis of the primary outcome measure, comparated to Impact of Weight on Quality Of Life at 12, 18 and 24 months. | 12, 18 and 24 month after surgery
  Impact of Weight on Quality Of Life : IWQOL It includes 36 items divided into five dimensions: physical, sexual, psychosocial,relationship with food, and experience of the diet.
  It allows us to assess the effects of dietary treatments on quality of life.. Each item is rated from 1 to 5, and each dimension is weighted to obtain a score out of 100. A high score indicates a good perceived quality of life related to obesity.

OTHER OUTCOMES:
Body schema measured at pre-surgical (M-6 and end of pre-operative course M-1) and post-surgical (M+12 and M+24) assessments. | at 6 and 1 month before surgery, and at 12, 18 and 24 months before surgery
  Body schema measured by SKIN. For each participant, an average difference between the perceived distance and the actual applied distance is calculated for each body part (thigh, abdomen, arm, shoulder (neutral zone)). A positive difference corresponds to an oversizing of the tactile surface of the body, while a negative difference corresponds to an undersizing of the tactile surface of the body
Body schema measured at pre-surgical (M-6 and end of pre-operative course M-1) and post-surgical (M+12 and M+24) assessments compared between the quality of life trajectory groups defined by the analysis of the primary judgment criterion | at 6 and 1 month before surgery, and at 12, 18 and 24 months before surgery
  Body schema measured by SKIN. For each participant, an average difference between the perceived distance and the actual applied distance is calculated for each body part (thigh, abdomen, arm, shoulder (neutral zone)). A positive difference corresponds to an oversizing of the tactile surface of the body, while a negative difference corresponds to an undersizing of the tactile surface of the body

CONTACTS AND LOCATIONS:
Overall Officials: Cécile BOSSU ESTOUR, Principal Investigator — CH Metropole Savoie
Locations (1):
- Centre Hospitalier Métropole Savoie, Chambéry, Savoie, France

IPD SHARING:
Plan to Share IPD: No